CLINICAL TRIAL: NCT00079716
Title: A Phase I, Multi-Dose Study of SGN-40 (Anti-huCD40 mAb) in Patients With Refractory or Recurrent Multiple Myeloma
Brief Title: Study of SGN-40 in Patients With Refractory or Recurrent Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Nancy Whiting, PharmD, Seattle Genetics, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG040-0001
Record Dates: First submitted 2004-03-11; First posted 2004-03-16 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Myeloma
Keywords: Antigens, CD40; Antibody, Monoclonal; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhagic Disorders; Hemostatic Disorders; Immunoproliferative Disorders; Lymphoproliferative Disorders; Paraproteinemias; Vascular Diseases; Antibody-Dependent Cell Cytotoxicity
MeSH Terms: conditions — Multiple Myeloma; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhagic Disorders; Hemostatic Disorders; Immunoproliferative Disorders; Lymphoproliferative Disorders; Paraproteinemias; Vascular Diseases | interventions — dacetuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SGN-40 (anti-huCD40 mAb)

INTERVENTIONS:
Drug: SGN-40 (anti-huCD40 mAb) — 0.5-8 mg/kg IV (in the vein) on Day 1; 0-8 mg/kg on Day 4; 0.5-16 mg/kg on Days 8 and 15; 0-16 mg/kg on Day 29.
  Other Names: dacetuzumab

SUMMARY:
The purpose of this study is to determine the safety and activity of SGN-40 in a weekly dosage schedule as a single agent.

DETAILED DESCRIPTION:
This is an open-label, multi-dose, single-arm, phase I, dose-escalation study to define the toxicity profile, maximum tolerated dose (MTD), pharmacokinetics, and antitumor activity of SGN-40 in patients with refractory or recurrent multiple myeloma.

A minimum of three patients will be entered into each dose-level cohort. All patients will receive a dose-loading schedule during the first two weeks. The maximum weekly dose will be 16mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have refractory or recurrent secretory multiple myeloma (MM).
2. Patients must have failed at least two different prior systemic therapies for MM.
3. Patients may have received a maximum of five cytotoxic regimens.
4. Patients who have received any of the following must complete within the specified time frame below:

   * Autologous stem cell transplant - 12 weeks prior to first dose
   * Nitrogen Mustard agents, Melphalan, BCNU, IVIG, or monoclonal antibody therapy - 6 weeks prior to first dose
   * Chemotherapy, Radiation, or other therapies for MM - 4 weeks prior to first dose
5. Patients who have not undergone autologous stem cell transplantation must be either ineligible for stem cell transplantation or, if eligible, must have refused treatment by autologous stem cell transplantation.
6. Patients must have an ECOG performance status of ≤ 2 and a life expectancy > three months.
7. Patients must be available for periodic blood sampling, study-related assessments, and management of toxicity at the treating institution for the entire duration of the study.
8. Patients must be at least 18 years of age.
9. Females of childbearing potential must have a negative β-HCG pregnancy test result within three days of enrollment. All patients must plan to use an effective contraceptive method during the course of the study.
10. Patients must meet baseline lab data requirements.
11. Patients must give written informed consent.

Exclusion Criteria:

1. Patients with non-secretory MM or solitary plasmacytoma or plasma cell leukemia.
2. Patients with a history of allogeneic transplantation.
3. Patients receiving plasmapheresis within four weeks prior to enrollment.
4. Patients undergoing major surgery within four weeks prior to enrollment.
5. Patients with a known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation.
6. Patients with a history of other malignancies during the past five years with the exception of adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ.
7. Patients with any active viral, bacterial, or systemic fungal infection within four weeks of enrollment.
8. Patients with a history of significant chronic or recurrent infections requiring treatment.
9. Patients with a history of active thrombosis within three months of enrollment.
10. Patients with a history of pulmonary embolism.
11. Patients with a history of migraines or severe headaches requiring medical therapy within 12 months of enrollment.
12. Patients who are pregnant or breastfeeding.
13. Patients with uncontrolled hypercalcemia.
14. Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment.
15. Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-03; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Adverse events and lab abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Whiting, PharmD, Study Director — Seagen Inc.
Locations (5):
- United States (5):
  - James R. Berenson M.D., Inc., West Hollywood, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cornell University, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Result] Hayashi T, Treon SP, Hideshima T, Tai YT, Akiyama M, Richardson P, Chauhan D, Grewal IS, Anderson KC. Recombinant humanized anti-CD40 monoclonal antibody triggers autologous antibody-dependent cell-mediated cytotoxicity against multiple myeloma cells. Br J Haematol. 2003 May;121(4):592-6. doi: 10.1046/j.1365-2141.2003.04322.x. PMID 12752100
- [Result] Hussein M, Berenson JR, Niesvizky R, Munshi N, Matous J, Sobecks R, Harrop K, Drachman JG, Whiting N. A phase I multidose study of dacetuzumab (SGN-40; humanized anti-CD40 monoclonal antibody) in patients with multiple myeloma. Haematologica. 2010 May;95(5):845-8. doi: 10.3324/haematol.2009.008003. Epub 2010 Feb 4. PMID 20133895
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20133895